CLINICAL TRIAL: NCT02617706
Title: A Prospective, Randomized, Parallel Study Comparing Transdermal, Continuous Oxygen Delivery to Standard of Care to Assess Postoperative Wound Infection Rate in Colon and Rectal Resections
Brief Title: Transdermal Continuous Oxygen Therapy for Infection Prophylaxis in High- Risk Patients Undergoing Colon Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: financial reasons
Sponsor: Neogenix, LLC dba Ogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPF-615
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2016-10

CONDITIONS: Anorectal Surgeries
Keywords: Anorectal surgeries; infection; topical oxygen
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal Continuous Oxygen Therapy (Experimental): EPIFLO® working study unit, all day, every day for 2 - 4 weeks + standard wound care
  Interventions: Device: Epiflo
- Standard of care (No Intervention): standard wound care for 4 weeks

INTERVENTIONS:
Device: Epiflo — Transdermal continuous oxygen therapy is oxygen delivery to the wound site directly. Ogenix makes a small portable oxygen concentrator (Trade Name: EPIFLO) that makes continuous transdermal delivery of oxygen possible. It is a 3 ounce oxygen generator that continuously delivers 3 ml of pure oxygen to the wound site.
  Other Names: TCOT, Transdermal Continuous Oxygen Therapy
  Arms: Transdermal Continuous Oxygen Therapy

SUMMARY:
EPIFLO® unit along with standard wound care vs only standard wound care for Surgical site infections (SSI).

DETAILED DESCRIPTION:
Anorectal procedures more often lead to surgical site infections. Such infections are unfortunately frequent and can be difficult for the patient and the treating physician. Wound hypoxia has been identified as a pathogenic mechanism behind wound infection and poor healing. Transdermal oxygen delivery (EPIFLO) is intended to promote the healing process in chronic wounds as an adjunct to standard wound care in wound management and treatment

ELIGIBILITY:
Inclusion Criteria:

* Elective colo-rectal surgery with or without anastomosis and with or without stoma
* Patient age: 18-80

Exclusion Criteria:

* Pregnancy

  * Anesthesiology ASA score of 4 or above
  * fever or existing signs of infection at the time of surgery
  * Diabetes Mellitus type I or II with HbA1C level 12% or more
  * Persons with decubitus or diabetic ulcers
  * Subjects with peritoneal metastases
  * Patients with severe malnutrition as indicated by Prealbumin value of <20
  * BMI ≥50

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with surgical site infections measured with the Southampton Scoring System. The number of subjects with infection of the surgical site will be compared using chi-square or Fisher Exact test. | 30 days
  The primary objective of this study is to assess surgical site infection within 30 days of surgery for "high risk" patients undergoing colo-rectal surgery in patients receiving adjunct Transdermal Continuous Oxygen therapy vs. standard of care control Measures as either yes infection or no infection

SECONDARY OUTCOMES:
Severity of infection measured with the Southampton Scoring System | 30 days
  Severity of infection using Southampton Scoring System. To maintain the trial-wise Type I error rate at 0.05, a closed test procedure will be used for the secondary endpoints
Number of days until patients surgical site is healed | 30 days
  Time to heal. To maintain the trial-wise Type I error rate at 0.05, a closed test procedure will be used for the secondary endpoints
Resource utilization - cost of treatments, hospital stays, bandages, nursing care | 30 days
  Resource utilization - cost of treatments, hospital stays, bandages, nursing care all measured in dollar amounts and then summed

CONTACTS AND LOCATIONS:
Overall Officials: Sarang Sarangapani, Ph.D., Study Director — Neogenix,LLC
Locations (1):
- Department of General Surgery Allegheny General Hospital, Pittsburgh, Pennsylvania, United States